CLINICAL TRIAL: NCT00778232
Title: A Relative Bioavailability Study of 800 mg Gabapentin Tablets Under Non-Fasting Conditions
Brief Title: Bioequivalence Study of Gabapentin 800 mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R01-826
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Gabapentin tablets 800 mg fed conditions
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Gabapentin tablets 800 mg by Ranbaxy Laboratories Limited
  Interventions: Drug: Gabapentin tablets 800 mg
- 2 (Active Comparator): Neurontin ® 800 mg tablets of Parke Davis Pharmaceuticals Ltd
  Interventions: Drug: Gabapentin tablets 800 mg

INTERVENTIONS:
Drug: Gabapentin tablets 800 mg

SUMMARY:
This study compared the relative bioavailability (rate and extent of absorption) of Gabapentin tablets 800 mg by Ranbaxy Laboratories Limited with that of Neurontin ® 800 mg tablets of Parke Davis Pharmaceuticals Ltd. Distributed by Parke-Davis, division of Warner-Lambert Co. following a single oral dose (1x800 mg tablet) in healthy adult volunteers under non-fasting conditions.

DETAILED DESCRIPTION:
A single oral dose of the test or the reference product was administered to 22 healthy adult human volunteers on two separate occasions under non-fasting conditions with at least a 7 day washout between the doses. Food and the fluid intake were controlled during each confinement period.

Twenty two (22) healthy adult human volunteers (12 males and 10 females) were enrolled in the study. All twenty two (22) subjects successfully completed the clinical portion of the study

ELIGIBILITY:
Inclusion Criteria:

1. All volunteers selected for the study will be healthy men or women 18 years of age or older at the time of dosing
2. The weight will no exceed ± 20% for the height and body frame as per desirable weight for adults - 1983 Metropolitan height and weight table
3. If female and Of Child bearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator (s), such as condoms , foams, jellies, diaphragm, intrauterine devices (IUD), or abstinence; or Is postmenopausal for at least 1 year; or Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

1. volunteers with a recent history of drug or alcohol addiction or abuse
2. Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system (s) or psychiatric disease (as determined by the clinical investigators)
3. Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant
4. Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen
5. Volunteers demonstrating a positive drug abuse screen when screened for this study
6. Female volunteers demonstrating a positive pregnancy screen
7. Female volunteers who are currently breast feeding
8. Volunteers with a history of allergic response (s) to Gabapentin or related drugs
9. Volunteers with a history of clinically significant allergies including drug allergies
10. Volunteers with a clinically significant illness during the 4 weeks prior to period I dosing (as determined by the clinical investigators)
11. Volunteers who are currently using tobacco products
12. Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to period I dosing
13. Volunteers who report donating greater than 150 mL of blood within 30 days prior to period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study
14. Volunteers who have donated plasma (eg. Plasmapheresis) within 14 days prior to period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study
15. Volunteers who report receiving any investigational drug within 30 days prior to period I dosing
16. Volunteers who report taking any systemic prescription medication in the 14 days prior to period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-10; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html